CLINICAL TRIAL: NCT05453539
Title: A Phase 1, Controlled, Open-label, Single Dose, Dose-escalation, Clinical Proof-of-concept Study of MRI Enhanced With ADx-001 (DSPE-DOTA-Gd Liposomal Injection) in Patients With Brain Amyloid Deposits as Demonstrated by Amyloid PET
Brief Title: Proof-of-concept Study of New Imaging Diagnostic in Patients With Suspected Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A temperature excursion occurred at the drug supplier's storage facility, which led to the loss of a significant portion of the IMP stock. Consequently, there is not enough IMP available to support continued recruitment
Sponsor: Alzeca Biosciences, Inc. (Industry)
Collaborators: pharmtrace klinische Entwicklung GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: ADx-001-101-POC; 2021-003399-14 (EudraCT Number)
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Healthy volunteers dose level 1 (Experimental): 0.53 mL ADx-001 / kg
  Interventions: Drug: DSPE-DOTA-Gd Liposomal Injection
- Patients dose level 1 (Experimental): 0.53 mL ADx-001 / kg
  Interventions: Drug: DSPE-DOTA-Gd Liposomal Injection
- Patients dose level 2 (Experimental): 1 mL ADx-001 / kg
  Interventions: Drug: DSPE-DOTA-Gd Liposomal Injection
- Patients dose level 3 (Experimental): 2 mL ADx-001 / kg
  Interventions: Drug: DSPE-DOTA-Gd Liposomal Injection
- Patients dose level 4 (Experimental): 4 mL ADx-001 / kg
  Interventions: Drug: DSPE-DOTA-Gd Liposomal Injection

INTERVENTIONS:
Drug: DSPE-DOTA-Gd Liposomal Injection — Single dose, intravenous infusion
  Other Names: ADx-001

SUMMARY:
This study is a Phase 1, first-in-human, multi-center study to establish safety of ADx-001 in healthy volunteers, and safety and proof of concept in patients with confirmed amyloid plaques in the brain (confirmed by amyloid positron emission tomography (PET)). ADx-001 is a novel, intravenously delivered, Gd- containing molecularly targeted liposomal product that is being developed for use in contrast-enabled MR imaging of amyloid plaques.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is an age-related neurodegenerative disorder of the brain and the most common cause of dementia. It is characterized by the development of amyloid plaques and neurofibrillary tangles. The A/T/N diagnostic criteria for AD, published by the National Institutes for Aging and the Alzheimer's Association (2018) identify amyloid plaques as a necessary condition for Alzheimer's disease.

Magnetic resonance imaging (MRI) is an essential neuroimaging examination for patients with Alzheimer's disease. MRI allows for the exclusion of other causes of dementia, such as normal pressure hydrocephalus, brain tumors, subdural hematoma, or cerebrovascular disease. MRI also permits the assessment of the atrophy pattern which may provide additional diagnostic or predictive information. To date, however, MRI cannot prove the existence of amyloid plaques in the brain.

Recently, amyloid-targeting radiopharmaceuticals have been approved by several Regulatory Authorities for use with Positron Emission Tomography (PET) imaging. Amyloid PET imaging is a sensitive imaging biomarker for Alzheimer's disease, but PET is associated with radiation exposure and has limited availability.

ADx-001 is a novel, intravenously delivered, macrocyclic gadolinium (Gd)-based molecularly targeted liposomal product that is being developed for use in contrast-enabled MR imaging of amyloid plaques. ADx-001-enabled MRI is expected to allow the detection of amyloid plaques in the human brain with sensitivity that is comparable to amyloid PET imaging.

This study is a Phase 1, first-in-human, study to collect safety data and obtain proof-of-concept of ADx-001 in healthy volunteers and subjects with proven amyloid plaques. Data from this study will be used to support future clinical studies with ADx-001 in AD patients.

. The study is designed in 2 parts. The first part in healthy volunteers is supposed to assess safety and tolerability in humans. In this study phase, 6 healthy volunteers will be included and receive a single dose of 0.016 mmol Gd/kg body weight, each. The first volunteer will be a sentinel and observed for 14 days before the next volunteers will be included. Volunteers will be recruited one-by-one with at least 24 h between the inclusion of subsequent volunteers.

The second part in patients with proven amyloid plaques (proven by amyloid PET) is supposed to provide proof of concept of ADx-001 MR signal enhancement in amyloid-rich brain regions and to identify the lowest ADx-001 dose able to delineate amyloid plaques in the human brain.

The patient part will use a dose escalation design with a maximum of 4 dose groups, with 3-6 patients in each dose group. The starting dose for the first dose level will be 0.016 mmol Gd/kg based on the NOAEL (0.5 mmol Gd/kg) established in the nonclinical development program, the safety factor of 0.1 and the human equivalent dose (HED) conversion factor of 0.32 (0.5 mmol Gd/kg x 0.1 x 0.32 = 0.016 mmol Gd/kg). Dose escalation will be based on findings in MRI and the occurrence of adverse events. Dose will be increased until no further increase in imaging signal is expected; stopping rules will define the stop of dose escalation (or the trial) based on safety considerations.

All study participants will need to be kept in-patient for observation for 72 hours after administration of ADx-001. At each dose level, the first patient will be a sentinel and followed for 14 days after the dose (or until early termination). If no clinically relevant adverse events or safety concerns occur during the first 14 days, additional 2 patients will be sequentially administered ADx-001 at the same dose with at least 24 h between the patients.

A Dosing Committee (DC) will oversee dose escalation of this trial. The DC will be composed of a board-certified radiologist, a physician specialized in a clinical discipline with experience in the administration of injectable liposome formulations, and a board-certified nuclear medicine physician as voting members. The DC will evaluate imaging and safety data, decide if further dose increases are expected to increase imaging signal, decide if the trial must be stopped following predefined stopping rules, decide if additional patients are to be included at a given dose level, and propose the next dose level. It is expected that dose levels will be gradually increased; however, the DC may also decide to lower the ADx-001 dose (especially after imaging of patients at the first dose if signal enhancement in amyloid plaques is already visible and judged as sufficient), or decide that no further dose levels are to be tested. The DC may also recommend different imaging time points (as long as the total number of imaging time points remains unaffected).

The following dose escalation criteria will be used:

* If no dose-limiting toxicity (DLT) has been seen in the first 3 subjects in a dose level and imaging signal is expected to increase with higher doses, then enrollment/dosing may move to the next higher dose level.
* If a DLT is seen in one of the first three subjects in a dose level, an additional 3 subjects will be enrolled into that same dose cohort. If only 1 DLT is seen in the first 6 subjects in a dose level and imaging signal is expected to increase with higher doses, then enrollment/dosing may move to the next higher dose level.
* Development of DLTs in 2 or more subjects in a specific dose cohort will indicate that the amount of drug tolerated has been exceeded, and further dose escalation will be terminated irrespective of imaging findings.
* The DC may recommend the next dose level be reduced from the previous dose (relevant for the first dose level in patients).

In all patients, amyloid PET imaging will serve as a comparator. Eligible patients will have a documented positive amyloid PET scan obtained within the 12 months prior to inclusion into this study and are able to provide the original DICOM images of the PET scan to the imaging core lab.

Patient recruitment will be done in a staggered approach. The time interval between injection with ADx-001 of the sentinel and subsequent patients is 14 days, at minimum. Safety follow-up of at least 7 days must be available in all 3 patients (or 6 patients if 1 DLT has been observed) of a dose level before the next higher dose level is started.

ELIGIBILITY:
Inclusion Criteria:

For healthy volunteers

1. 50-75 years old (inclusive)
2. Women of child-bearing potential must have a negative serum pregnancy test and agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of the study and for 3 months after completion of dosing; men enrolled on this protocol must agree to use adequate contraception prior to study entry, for the duration of the study and for 3 months after completion of dosing; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
3. Signed informed consent prior to any study specific tests or procedures
4. Healthy, based on medical history, physical examination, electrocardiogram (ECG), and laboratory tests

For patients with amyloid plaques in PET:

1. 59-85 years old inclusive
2. Proven amyloid deposits in brain (amyloid PET)
3. Women of child-bearing potential must have a negative serum pregnancy test and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of the study and for 3 months after completion of dosing. Men enrolled on this protocol must agree to use adequate contraception prior to study entry and for 3 months after completion of dosing; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
4. Willing and able to provide written informed consent
5. The ability to provide consent determined and documented by a neurologist or psychiatrist.

Exclusion Criteria:

For healthy volunteers

1. Disturbances in fat metabolism [hyperlipemia, hyperlipoproteinemia or hypercholesterolemia (total cholesterol >260 mg/dL)]
2. History of allergic reactions attributed to any of the components of ADx-001, liposomes, other gadolinium contrast agents, or any other component of the formulation
3. Pathological liver function:

   1. Bilirubin > upper limit of normal, and/or
   2. AST (SGOT), ALT (SGPT) and Alkaline phosphatase > upper limit of normal
4. Calculated creatinine clearance < 60 mL/min/1.73 m2 (CKD-EPI formula)
5. Heart rate at rest <50 or >90 bpm
6. Systolic blood pressure <100 or >140 mmHg
7. Diastolic blood pressure <50 or >90 mmHg
8. Clinically relevant ECG findings, e.g., PQ >220 ms, QTc >450 ms, QRS >120 ms, branch bundle block, any sign of coronary heart disease
9. Unwillingness or inability to comply with procedures required in this protocol
10. Subjects who are currently receiving any other investigational agent, or who have received an investigational agent within the last 10 half-lives of the investigational agent
11. Having tested positive for COVID-19 within 4 weeks of inclusion
12. Any known disposition for allergic, anaphylactoid, hypersensitivity or idiosyncratic reactions, e.g. any history of clinical signs of hypersensitivity reaction to any agent (including, but not limited to, any allergen, food, drug, chemical, or contrast agent)
13. Use of systemic or topically active medication or herbal remedies, prescription or non-prescription, from screening to the first drug administration. Only use of contraceptives and occasional use of paracetamol, aspirin, or ibuprofen is permissible.
14. Any severe disease within the last 4 weeks prior to the first study drug administration
15. Any malignant tumor and history thereof within last 5 years
16. Any other medical condition which, at the discretion of the investigator, would make study participation unadvisable
17. Any clinically relevant finding at the physical examination
18. Blood donation or plasmapheresis within 4 weeks prior to screening
19. Women of child-bearing potential: pregnancy, positive pregnancy test, or lactation
20. Positive human immunodeficiency virus antibodies (HIV-1/2 Ab), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibody (HCV-Ab) tests
21. Regular alcohol consumption equivalent to >20 g alcohol per day
22. Urine screen positive for any drug
23. Positive alcohol breath test
24. Subject is in custody by order of an authority or a court of law
25. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site) or employee of the sponsor
26. Criteria which, in the opinion of the investigator, preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety

For patients with amyloid plaques in PET:

1. Disturbances in fat metabolism [hyperlipemia, hyperlipoproteinemia or hypercholesterolemia (total cholesterol >260 mg/dL)]
2. History of allergic reactions attributed to any of the components of ADx-001, liposomes, other gadolinium contrast agents, or any other component of the formulation
3. Patients with history of cancer treatment in the last 6 months or currently receiving cancer treatment
4. Major surgery within four weeks prior to Screening
5. History or presence of a neurological or psychiatric diagnosis other than AD (not limited to but including for example, stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, major depression, brain tumors, etc.) that in the opinion of the investigator may limit compliance with study requirements, or compromise protocol objectives in the opinion of the investigator and/or the sponsor
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or compromise protocol objectives in the opinion of the investigator and/or the sponsor
7. Unwillingness or inability to comply with procedures required in this protocol
8. Patients who are currently receiving any other investigational agent, or who have received an investigational agent within the last 10 half-lives of the investigational agent
9. Inability to undergo MRI
10. Pathological coagulation status (PT-INR/PTT >1.5 times the upper limit of normal)
11. Pathological hematologic status:

    * Granulocyte < 1500 cells/mm3, and/or
    * Platelet count < 150,000 (plt/mm3), and/or
    * Hemoglobin < 10 g/dL
12. Pathological liver function:

    * Bilirubin > upper limit of normal, and/or
    * AST (SGOT), ALT (SGPT) and Alkaline phosphatase > upper limit of normal
13. Calculated creatinine clearance < 60 mL/min/1.73 m2 (CKD-EPI formula)
14. Cannot tolerate the recommended pretreatment
15. Having tested positive for COVID-19 within 4 weeks of inclusion

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 0-28

SECONDARY OUTCOMES:
The number of brain regions identified the same way in ADx-001 enhanced MRI and in amyloid-PET | Screening - day 4
The amount of contrast enhancement in the amyloid positive brain regions in different dose levels | Screening - day 4

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Stoecklein, Principal Investigator — LMU Klinikum
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - LMU Klinikum, Munich

IPD SHARING:
Plan to Share IPD: No